CLINICAL TRIAL: NCT00778193
Title: A Randomized, Blinded, Placebo-Controlled Study of the Effect of Naproxen, Aspirin, Celecoxib, or Clopidogrel on Gastroduodenal Healing
Brief Title: Effect of Naproxen, Aspirin, Celecoxib, or Clopidogrel on the Healing of Stomach and Intestinal Ulcers
Acronym: Lesions2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Associates of New York, LLP (Other)
Responsible Party: James Asienberg, MD, Research Associates of New York
Other Study IDs: Healing Study; GA319181
Record Dates: First submitted 2008-07-24; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Gastroduodenal Ulcer
Keywords: NSAID; ulcer; gastroduodenal ulcer; naproxen; aspirin; ASA; celecoxib; clopidogrel; healing; Cyclooxygenase 2 Inhibitors; Anti-Inflammatory Agents, Non-Steroidal; Platelet Aggregation Inhibitors; Wound Healing
MeSH Terms: conditions — Peptic Ulcer; Ulcer | interventions — Naproxen; Aspirin; Celecoxib; Clopidogrel; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- Aspirin (Experimental)
  Interventions: Drug: Aspirin
- Clopidogrel (Experimental)
  Interventions: Drug: Clopidogrel
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Naproxen — 1 tablet 500mg BID for 8 days
  Other Names: naprosyn; naproxen sodium; Aleve; Anaprox; Miranax; Naprogesic; Naprelan; Proxen; Synflex
  Arms: Naproxen
Drug: Aspirin — 1 tablet 81mg QD for 8 days
  Other Names: ASA; Bayer
  Arms: Aspirin
Drug: Celecoxib — 1 capsule 200mg QD for 8 days
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Clopidogrel — Day 0: 4 tablets QD for 1 day; Days 1-7: 1 tablet QD for 7 days
  Other Names: Plavix
  Arms: Clopidogrel
Drug: Placebo — 1 capsule BID for 8 days
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Gastroduodenal ulcers are extremely common in the community today. Though much has been written and observed concerning how ulcers form, not much has been described in the human model concerning how these ulcers heal. As numerous patients already suffer from gastrointestinal ulcers, further clarification of ulcer healing would be valuable in the treatment and management of these patients. The goal of this study is to investigate the effects of naproxen, aspirin, celecoxib, and clopidogrel on biopsy-induced gastroduodenal lesions in order to elucidate the mechanisms of ulcer healing. This single site, single-blind, randomized, placebo-controlled, one-week prospective study will examine ulcer healing through endoscopic, immunohistologic, and molecular PCR modalities.

DETAILED DESCRIPTION:
In order to assess the extent of healing of the biopsy sites, a 12-point scale was developed and validated.

After all of the procedures were complete, this scale was used to measure the effects of the study drugs on the healing of the biopsy-induced ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18-75
* Use of appropriate form of birth control for women of childbearing potential.

Exclusion Criteria:

* H pylori infection
* Use of NSAIDs within 2 weeks prior to start of enrollment
* Use of antacids or H-2 blockers within 2 weeks of enrollment
* Use of PPIs within 30 days of enrollment
* Corticosteroid use within 60 days of enrollment
* History of a previous ulcer
* Diagnosis of a bleeding diathesis or use of warfarin within 60 days of enrollment
* Use of cigarettes within 6 months of enrollment
* Consumption of >3 alcoholic beverages per day
* Hypersensitivity or allergy to NSAIDs, clopidogrel, or corn starch, or any contraindications to ingesting those substances
* The presence of an ulcer at a baseline endoscopy
* Endoscopically severe gastritis or duodenitis baseline endoscopy
* Moderate or severe inflammation located within the duodenal bulb or within 2cm of the pyloric channel at a baseline endoscopy
* Any gastroduodenal tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Aisenberg, MD, Principal Investigator — Research Associates of New York
Locations (1):
- Research Associates of New York, New York, New York, United States

REFERENCES:
- [Background] Desai JC, Sanyal SM, Goo T, Benson AA, Bodian CA, Miller KM, Cohen LB, Aisenberg J. Primary prevention of adverse gastroduodenal effects from short-term use of non-steroidal anti-inflammatory drugs by omeprazole 20 mg in healthy subjects: a randomized, double-blind, placebo-controlled study. Dig Dis Sci. 2008 Aug;53(8):2059-65. doi: 10.1007/s10620-007-0127-4. Epub 2008 Jan 26. PMID 18224442